CLINICAL TRIAL: NCT03631251
Title: Enhancing Analgesia With Non-Deceptive Placebos: A Proof-Of-Concept Pilot Study
Brief Title: Using Honest Placebos to Improve Pain Management in Hand Surgery Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Michael Bernstein, Postdoctoral Fellow, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000556
Record Dates: First submitted 2018-07-26; First posted 2018-08-15 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Hand or Wrist Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Placebo (Experimental): Open placebo in addition to the standard course of opioids. Opioids are given consistent with standard care.
  Interventions: Drug: Open Placebo

INTERVENTIONS:
Drug: Open Placebo — Open placebo in addition to the standard course of opioids. Opioids are given consistent with standard care.

SUMMARY:
America is in the midst of an opioid epidemic. One of the reasons opioid addiction and overdose deaths have recently increased is that doctors are frequently prescribing opioid medication as a treatment for pain. If it is possible to develop new ways of increasing the pain-relief patients experience from a set amount of opioids, then doctors might ultimately be able to prescribe fewer opioid medications, which could help curb the opioid crisis.

Although "placebos," a medication whose benefit derives solely from positive psychological factors rather than pharmacological factors, are often disparaged in medicine, research suggests that placebos can actually help reduce pain. In fact, there is reason to think that placebos are effective even when a patient knows they are taking a placebo.

The goal of the proposed study is to examine the feasibility of using an honest placebo to relieve pain for up to 20 real patients. People who are undergoing hand or wrist surgery or enrolled for upper extremity trauma in the Emergency Department and agree to participate will be asked to take placebo pills in addition to their standard course of opioid pills, given as part of standard care. Patients will also answer a few short questions over the phone once per day for seven days, and be invited to participate in an exit questionnaire at the end of the study. The investigators hypothesize that: 1) At least 50% of eligible participants will agree to enroll, 2) At least 80% of participants who are enrolled will be retained, and 3) Participants who are enrolled will take a placebo at least 50% of the time they also take an opioid pill

ELIGIBILITY:
Inclusion Criteria, University Orthopedics & Department of Plastic & Reconstructive Surgery:

* 18 years or older
* English Speaking
* Have a working phone
* Scheduled for hand or wrist surgery
* Able to provide informed consent Inclusion Criteria, Miriam Hospital Emergency Department
* 18 years or older
* English Speaking
* Have a working phone
* Able to provide informed consent
* Present for upper extremity trauma
* Are expected to be prescribed opioids at discharge
* Are expected to be discharged from the Emergency Department

Exclusion Criteria, University Orthopedics & Department of Plastic & Reconstructive Surgery::

* Known history of Substance Use Disorder
* Chronic pain
* Chronic opioid use
* The prescribing physician deems opioid medication not appropriate as part of standard care for any reason Exclusion Criteria, Miriam Hospital Emergency Department
* Known history of Substance Use Disorder
* Chronic pain
* Chronic opioid use
* Unlikely to follow-up (discretion of investigator and treating provider)
* Likely to receive surgical repair of the indicated injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Enrollment Percentage | Through study enrollment, 1 day
  Percentage of Eligible Patients who Enroll
Retention Rate | through study completion, approximately 2 months
  Percentage of Patients who are Retained at follow-up
Placebo Intake | 7 days
  Number of Placebos Participants Take
Placebo Analgesia | 7 days
  Analgesia associated with placebo pills

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University Orthopedics, East Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No